CLINICAL TRIAL: NCT05129514
Title: Imaging Lymphatic/CSF Drainage From the Head and Neck in Persons With Traumatic Brain Injury: Demonstration of Feasibility and Evaluation of Manual Therapy to Improve Drainage and Facilitate Cognitive Recovery
Brief Title: Imaging Lymphatic/Cerebrospinal Fluid (CSF) Drainage From the Head and Neck in Persons With Traumatic Brain Injury: Demonstration of Feasibility and Evaluation of Manual Therapy to Improve Drainage and Facilitate Cognitive Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: HeadStrong Foundation (Unknown)
Responsible Party: Principal Investigator, Eva Sevick, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0080
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Trauma, Brain; Neuroinflammation
Keywords: traumatic brain injury; lymphatic drainage; cerebrospinal fluid
MeSH Terms: conditions — Brain Injuries, Traumatic; Neuroinflammatory Diseases | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual Lymphatic Drainage (MLD) (Experimental)
  Interventions: Other: Manual Lymphatic Drainage (MLD)

INTERVENTIONS:
Other: Manual Lymphatic Drainage (MLD) — The participant will be placed in a supine position and manual lymphatic drainage will be performed for 50 minutes. During the three intervening days, daily 50 minute sessions of manual lymphatic drainage will be provided.

SUMMARY:
The purpose of this study is to determine whether a course of daily manual lymphatic drainage over the course of 5 days can improve lymphatic drainage function and cognitive outcomes and to determine whether single sessions of manual lymphatic drainage improves lymphatic drainage in moderate to severe traumatic brain injury (TBI) patients.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must complete the Female Enrollment Form. Those subjects of childbearing potential must have a negative urine pregnancy within 36 hours of study drug administration and also agree to use one of the medically accepted methods of contraception listed on the form for a period of one month following the study. Female subjects of non-childbearing potential, defined as physiologically incapable of becoming pregnant, must meet the criteria listed on the Female Enrollment form, but are not restricted to the use of contraception following study participation.
* Participants must be able to sit upright for periods of 30 minutes.
* Participants should have a body mass index between 19 and 30 kg/m2
* Initial post-resuscitation Glasgow Coma Scale score following blunt head trauma of 3 to 12 or coma (not due to sedation) greater than 6 hours. Emergence from Post-traumatic Amnesia as documented by serial administration of the Orientation-Log or Galveston Orientation and Amnesia Test
* Have an anticipated hospital length of stay of 5 days or more following screening and consent.
* Able to provide consent.

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Persons who are known to be allergic to iodine
* Persons who have extensive soft tissue damage to the neck region, including carotid artery dissection, spinal cord injury, or other conditions, that makes lymphatic drainage techniques undesirable.
* Women who are of child bearing potential who do not agree to use medically acceptable contraceptives for one month following the study.
* Subjects who are participating in another interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
change in Near-Infrared Fluorescence Lymphatic Imaging (NIRF-LI) assessment of lymphatic drainage | day 1, day 5
  2 NIRF-LI sessions will be conducted separated by 3 days.
change in cognitive test results as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)-Global health( GH) scale | day1,day2,day3,day4,day5
  Nine of the 10 PROMIS GH items are scored on a Likert scale from 1 to 5, with 5 representing the best health. Pain which is the 10th question is scored from 0(no pain) to 10(worst imaginable pain).
change in cognitive test results as assessed by the Patient Health Questionnaire-9 (PHQ-9) | day1,day2,day3,day4,day5
  This scale consists of a set of 9 questions each scored form 0(not at all) to 3 (nearly every day), a higher score indicating a worse outcome. Total score ranges form 0-27.
change in cognitive test results as assessed by the Multilingual Aphasia Examination III-Controlled Oral Word Association | day1,day2,day3,day4,day5
  This is used to asses phonemic fluency. Participant is asked to name words that begin with a particular letter in one minute and examiner will write down the words said by the participant. This will be reported y the number of words participants say in one minute
change in cognitive test results as assessed by the Trail Making Test(TMT) | day1,day2,day3,day4,day5
  Scores are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
change in cognitive test results as assessed by the learning trial | day1,day2,day3,day4,day5
  This will be assessed by the number of words participants can remember
change in cognitive test results as assessed by the delayed recall trial instructions | day1,day2,day3,day4,day5
  This will be assessed by the number of words participants can remember after 20-25 minutes delay
change in cognitive test results as assessed by the Semantic Category learning trial | day1,day2,day3,day4,day5
  There are 12 words that participants will categories as Four-legged Animals, precious stones and human dwellings for a total score from 0-12 a higher number indicates a better outcome
Change in processing speed, as assessed by the Wechsler Adult Intelligence Scale -IV | day1,day2,day3,day4,day5
  Two subtests from the Wechsler Adult Intelligence Scale - IV are used (Coding and Symbol Search). Age-adjusted standard scores are calculated for each of subtest. The 2 subtest scores are then combined to create the Processing Speed Index. Processing Speed Index will be reported as a percentile (0% to 100%), with a higher percentile indicating a better outcome

SECONDARY OUTCOMES:
Change in NIRF-LI detected lymphatic drainage | day1,day5
  response of NIRF-LI detected lymphatic drainage in response to manual lymphatic drainage by imaging drainage before and after manual lymphatic drainage

CONTACTS AND LOCATIONS:
Overall Officials: Eva Sevick, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No